CLINICAL TRIAL: NCT05971368
Title: A Comparative Study Between Ultrasound Guided Thoracic Paravertebral Block VS Ultrasound Guided Serrartus Anterior Muscle Block in Video-assisted Thoracoscopic Surgeries.
Brief Title: A Comparative Study Between Ultrasound Guided Thoracic Paravertebral Block VS Serrartus Anterior Muscle Block in VATS as Regard Their Effectiveness in Post-operative Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: paravertebral vs serratus
Record Dates: First submitted 2023-06-16; First posted 2023-08-02 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-06

CONDITIONS: Post Operative Pain, Acute
Keywords: regional anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Masking Description: * Group A: Patients will receive ultrasound guided thoraxic paravertebral block with 0.25% bupivacaine 0.4 ml/kg (max. 40 ml and not exceeding toxic dose of bupivacaine 2.5mg/kg) after induction of anesthesia.
  * Group B: Patients will receive ultrasound guided serratus anterior muscle block with 0.25% bupivacaine 0.4 ml/kg (max. 40 ml and not exceeding toxic dose of bupivacaine 2.5mg/kg) after induction of anesthesia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Patients will receive ultrasound guided thoracic paravertebral block (Active Comparator): Group A: Patients will receive ultrasound guided thoraxic paravertebral block with 0.25% bupivacaine 0.4 ml/kg (max. 40 ml and not exceeding toxic dose of bupivacaine 2.5mg/kg) after induction of anesthesia.
  Interventions: Procedure: thoracic paravertebal block
- Group B: Patients will receive ultrasound guided serratus anterior muscle block (Active Comparator): Group B: Patients will receive ultrasound guided serratus anterior muscle block with 0.25% bupivacaine 0.4 ml/kg (max. 40 ml and not exceeding toxic dose of bupivacaine 2.5mg/kg) after induction of anesthesia.
  Interventions: Procedure: serratus anterior muscle block

INTERVENTIONS:
Procedure: thoracic paravertebal block — o Group A: Patients will receive ultrasound guided thoraxic paravertebral block with 0.25% bupivacaine 0.4 ml/kg (max. 40 ml and not exceeding toxic dose of bupivacaine 2.5mg/kg) after induction of anesthesia.
  A high-frequency linear ultrasound probe will be placed between transverse processes from the T4 level (the level of port introduction) in the paramedian plane while patients is in the lateral decubitus position. The transverse processes, superior costotransverse ligaments, and pleura will be well visualized. The block needle (22 gauge) will be advanced until it crosses the superior costotransverse ligament. The prepared 0.25% bupivacaine will be administered at 0.4 mL/kg (max. 40 mL) in the thoracic paravertebral space. Depression of the pleura will be observed as a result of the spread of local anesthetic.
  Arms: Group A: Patients will receive ultrasound guided thoracic paravertebral block
Procedure: serratus anterior muscle block — Group B: Patients will receive ultrasound guided serratus anterior muscle block with 0.25% bupivacaine 0.4 ml/kg (max. 40 ml and not exceeding toxic dose of bupivacaine 2.5mg/kg) after induction of anesthesia.
  While the patient is in the supine position, a high-frequency linear ultrasound probe will be placed horizontally on the mid-axillary line at the level of 4th or 5th ribs on the side of the block. The serratus anterior, latissimus dorsi, and intercostal muscles will be identified. The block needle (22-gauge) will be advanced below the serratus anterior muscle (SAM) towards the fifth rib (using in-plane technique). The prepared 0.25% bupivacaine will be administered at 0.4 mL/kg (max. 40 mL) between the SAM and the rib. It will be observed that the solution of local anesthesia will spread between the SAM and the rib.
  Arms: Group B: Patients will receive ultrasound guided serratus anterior muscle block

SUMMARY:
A comparative study between ultrasound guided thoracic paravertebral block VS ultrasound guided serrartus anterior muscle block in video-assisted thoracoscopic surgeries as regard their effectiveness in post-operative analgesia

DETAILED DESCRIPTION:
The use of loco-regional analgesia is recommended to control postoperative pain after VATS as it allows opioid sparing and facilitates early postoperative rehabilitation. Different loco-regional analgesic techniques could be used to control pain after thoracic surgery such as a paravertebral block, an intercostal block and serratus plane block. In this study, Thoracic paravertebral nerve block will be compared to Serratus anterior nerve block, both will be done Ultrasound guided (USG) using bupivacaine (0.25%) for postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients American Society of Anesthesiologists physical status (ASA) I to II
* Both sexes.
* Aged ≥ 20 to ≤ 65years.
* Scheduled for VATS under general anesthesia.

Exclusion Criteria:

* Patient's refusal.
* Patients American Society of Anesthesiologists physical status (ASA) III to IV
* Patients with major spine deformities.
* Disruption of the local anatomy, secondary, for instance, to the presence of chest drains or surgical emphysema, resulting in difficulty in ultrasound interpretation and distortion of tissue planes.
* Patients with bleeding disorders and coagulopathy.
* Infection at the injection site.
* Known allergy to local anesthetics.
* Patients with pre-existing myopathy or neuropathy.
* Ipsilateral diaphragmatic paresis.
* Tumors in the paravertebral space at the level of injection.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-04 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
total amount of opioid consumption in the two groups according to change in VAS score | the first 24 hours postoperatively
  Postoperative pain will be assessed at time of evaluation or at any time the patient is complaining of pain by using visual analog scale (VAS) and VAS more than 3 will be managed by injection of nalbuphine 0.05mg / kg intravenously as a first rescue analgesia to reduce VAS score ≤ 3 and another titrating dose (2-3 mg nalbuphine) will be considered if the patient is still complaining in order to reach VAS score ≤ 3 (with maximum dose of 10 mg nalbuphine at a time)
visual analog scale (VAS) | the first 24 hours postoperatively
  Postoperative pain will be assessed at time of evaluation or at any time the patient is complaining of pain by using visual analog scale (VAS) and VAS more than 4 will be managed by injection of nalbuphine 5mg intravenously as a first rescue analgesia to reduce VAS score ≤ 3

SECONDARY OUTCOMES:
The onset of 1st analgesic request | The first 24 hours postoperatively
  Postoperative pain will be assessed by using visual analog scale (VAS) and VAS more than 4 will be managed by injection of nalbuphine 5mg intravenously as a first rescue analgesia to reduce VAS score ≤ 3. comparison will be done between the two groups in the onset of 1st analgesic request
mean arterial blood pressure of the patients | first 24 hours postoperatively
  After surgery, Patients will be observed immediately post-operative at 0 (PACU), and 2, 4, 8, 12, 24 hours after surgery for post-operative pain in form of increasing mean arterial blood pressure as a sign of uncontrolled pain
onset of ambulation | first 24 hours postoperatively
  controlling pain postoperatively will help in early ambulation which is a major goal post operative to decrease complications
complication of nerve block | first 24 hours postoperatively
  as hematoma , infection , pneumothorax .
heart rate of the patients | first 24 hours postoperatively
  After surgery, Patients will be observed immediately post-operative at 0 (PACU), and 2, 4, 8, 12, 24 hours after surgery for post-operative pain in form of increasing heart rate above 90 (pulse per min )as a sign of uncontrolled pain

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Ain shams university, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided